CLINICAL TRIAL: NCT05203588
Title: The Effects of Denosumab on Bone Fusion and Bone Metabolism in Osteoporotic Patients With Lumbar Degenerative Disease After Lumbar Interbody Fusion
Brief Title: Effects of Denosumab on Bone Fusion in Osteoporotic Patients After Lumbar Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021SL031
Record Dates: First submitted 2021-12-08; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Osteoporosis; Fusion of Spine, Lumbar Region
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Patients in this group are received denosumab (60 mg) subcutaneously at one week and 26 weeks after the lumbar fusion surgery, combined with receiving daily calcium (≥1·0 g) and vitamin D (≥400 IU).
  Interventions: Drug: Denosumab 60 mg/ml Injectable Solution [Prolia]; Drug: calcium and vitamin D
- Control group (Sham Comparator): Patients in this group are only received daily calcium (≥1·0 g) and vitamin D (≥400 IU) after the lumbar fusion surgery.
  Interventions: Drug: calcium and vitamin D

INTERVENTIONS:
Drug: Denosumab 60 mg/ml Injectable Solution [Prolia] — Denosumab, 60mg(1ml), subcutaneously, totally two times, with one time at 1-week postoperatively and another time at 26-week postoperatively.
  Arms: Experimental group
Drug: calcium and vitamin D — calcium (≥1·0 g) and vitamin D (≥400 IU).

SUMMARY:
Lumbar fusion is an accepted and effective technique for the treatment of lumbar degenerative disease. As the population ages, disability associated with spinal pathology and spinal surgery is rapidly increasing and there is a concomitant increase in prevalence of osteoporosis which is a detrimental factor for Lumbar fusion and instrumentation. Osteoporosis-related bone fragility is a primary reason for spinal fusion failure, implant fixation failure, and vertebral compression fractures above or below the fusion sites.

Denosumab is a human monoclonal antibody against RANKL, it inhibits osteoclast mediated bone destruction and has been found to be effective in treating osteoporosis, including reducing bone turnover markers, increasing bone mineral density (BMD), and reducing fractures. But few studies focus on the effects of Denosumab on lumbar fusion. In this study, we include osteoporotic patients with lumbar degenerative disease who have had lumbar interbody fusion surgery. The patients were randomized to either treatment of Denosumab or no treatment. All these patients are followed at 3, 6, 9, 12 months postoperation. During these periods, we detect bone metabolism and bone fusion of these patients. Finally, we would report whether Denosumab can improve bone metabolism and promote bone fusion or not.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of degenerative lumbar diseases with symptoms of low-back pain and/or leg pain for at least 3 months, which was not be adequately controlled by nonoperative treatments.
2. Diagnosis of osteoporosis, defined as a bone mineral density (BMD) at lumbar or femoral neck with 2.5 standard deviations or more below the mean peak bone mass (T scores <-2.5 SD) measured by dual-energy X-ray absorptiometry (DXA).
3. Patients will be underwent single-level or two-level lumbar interbody fusion.

Exclusion Criteria:

1. Paget disease of bone,
2. Low laboratory tests for calcium,
3. Previous radiation treatment or fusion surgery to lumbar spine,
4. Bone tumors,
5. Bone infection,
6. Acute vertebral fractures
7. Severe spinal deformities such as degenerative scoliosis,
8. Other metabolic bone disease,
9. History of a anti-osteoporosis medication
10. Combined with severe morbidities,
11. Uncorrected bleeding diatheses
12. Application of steroids.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
lumbar fusion rate | 3-month post-operation
  Fusion rate assessed by CT scan and dynamic radiograph
lumbar fusion rate | 6-month post-operation
  Fusion rate assessed by CT scan and dynamic radiograph
lumbar fusion rate | 9-month post-operation
  Fusion rate assessed by CT scan and dynamic radiograph
lumbar fusion rate | 12-month post-operation
  Fusion rate assessed by CT scan and dynamic radiograph

SECONDARY OUTCOMES:
Bone metabolic markers including serum carboxy terminal cross-linked telopeptide of type I collagen (β-CTX) and osteocalcin (OCN) | pre-operation
  To assess bone metabolism, serum samples will be collected under nonfasting conditions, and the concentrations of β-CTX) and osteocalcin (OCN) will be measured using ELISA as biomarkers of bone resorption and formation, respectively.
Bone metabolic markers including serum carboxy terminal cross-linked telopeptide of type I collagen (β-CTX) and osteocalcin (OCN) | 3-month post-operation
  To assess bone metabolism, serum samples will be collected before and after surgery under nonfasting conditions, and the concentrations of β-CTX) and osteocalcin (OCN) will be measured using ELISA as biomarkers of bone resorption and formation, respectively.
Bone metabolic markers including serum carboxy terminal cross-linked telopeptide of type I collagen (β-CTX) and osteocalcin (OCN) | 6-month post-operation
  To assess bone metabolism, serum samples will be collected before and after surgery under nonfasting conditions, and the concentrations of β-CTX) and osteocalcin (OCN) will be measured using ELISA as biomarkers of bone resorption and formation, respectively.
Bone metabolic markers including serum carboxy terminal cross-linked telopeptide of type I collagen (β-CTX) and osteocalcin (OCN) | 9-month post-operation
  To assess bone metabolism, serum samples will be collected before and after surgery under nonfasting conditions, and the concentrations of β-CTX) and osteocalcin (OCN) will be measured using ELISA as biomarkers of bone resorption and formation, respectively.
Bone metabolic markers including serum carboxy terminal cross-linked telopeptide of type I collagen (β-CTX) and osteocalcin (OCN) | 12-month post-operation
  To assess bone metabolism, serum samples will be collected before and after surgery under nonfasting conditions, and the concentrations of β-CTX) and osteocalcin (OCN) will be measured using ELISA as biomarkers of bone resorption and formation, respectively.

OTHER OUTCOMES:
Bone mineral density (BMD) | Pre-operation
  BMD will be measured at the lumbar spine or femoral neck by DXA before surgery.
Bone mineral density (BMD) | 6-month post-operation
  Due to instrumentation at the lumbar site, BMD will be measured only at the femoral neck by DXA after surgery.
Bone mineral density (BMD) | 12-month post-operation
  Due to instrumentation at the lumbar site, BMD will be measured only at the femoral neck by DXA after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Changgui Shi, M.D., Principal Investigator — Shanghai changzheng hospital, Naval Medical University
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No